CLINICAL TRIAL: NCT00719446
Title: Patient Outcomes 6 and 12 Months After ALTA, OMEGA, EDEN and SAILS ARDS Network Trials
Brief Title: Evaluating Health Outcomes and QOL After ALI Among Participants of the ALTA, OMEGA, EDEN, and SAILS ARDS Network Trials
Acronym: ALTOS
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Dale Needham, Associate Professor, Johns Hopkins University
Other Study IDs: 589; R01HL091760 (NIH)
Record Dates: First submitted 2008-07-18; First posted 2008-07-21 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Respiratory Distress Syndrome, Adult
Keywords: Acute Lung Injury
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Acute lung injury (ALI) is a severe lung condition that causes respiratory failure. The ARDS Network (ARDSNet) is a National Heart, Lung, and Blood Institute-sponsored network that is focused on improving treatments for people with ALI and a similar condition called acute respiratory distress syndrome (ARDS). This study will evaluate participants who were enrolled in one of three ARDSNet studies to examine how the treatments carried out in the prior studies affect participants' long-term health outcomes and quality of life.

DETAILED DESCRIPTION:
ALI, a life-threatening condition that involves inflammation of the lungs and fluid accumulation in the air sacs, typically leads to low blood oxygen levels and respiratory failure. Common causes of ALI include pneumonia, sepsis, and lung trauma. Symptoms, including breathing difficulty, low blood pressure, and organ failure, usually develop within 24 to 48 hours of the original injury or illness. Most patients require immediate care in an intensive care unit (ICU), and the main form of treatment is mechanical ventilation, which delivers oxygen and a continuous level of pressure to the damaged lungs. The ARDS Network (ARDSNet) is a group of hospitals and medical centers that conduct research to improve treatment options for people with ARDS and ALI. This study will enroll people who participated in the ARDSNet's ALTA, OMEGA, EDEN, or SAILS study; these studies are investigating new treatments to improve survival and reduce the amount of time people remain on mechanical ventilation in the ICU after ALI. It is not known whether the ARDSNet's treatments have any prolonged benefit for patients after they leave the hospital. The purpose of this study is to evaluate participants' quality of life and long-term health outcomes after they receive the ALTA, OMEGA, EDEN, or SAILS study treatments.

This study will enroll participants who were in the ALTA, OMEGA, EDEN, or SAILS study. ARDS Network trial participants from sites that approved this follow-up study will be contacted by phone at 6 and 12 months to complete a collection of surveys. These surveys assess quality of life, mental health, memory and cognition, physical functioning, fatigue, employment and health insurance status, and health care utilization. At the end of each follow-up, participants will be asked for feedback regarding their experience during the follow-up.

For participants from a sub-set of ARDS Network study sites participating in this study, researchers will review participants' medical records and information collected during the ARDSNet studies. Six and 12 months after ALI, participants will attend study visits at which time walking ability, lung function, and muscle strength will be measured. Weight, dietary changes, and changes in muscle and fat composition will also be assessed. Participants will take part in interviews to evaluate memory and cognition. If participants cannot attend the study visits, research staff will either visit participants' homes to complete the evaluations or conduct some of the evaluations over the phone.

ELIGIBILITY:
Inclusion Criteria:

* Participated in the ALTA, EDEN, OMEGA, or SAILS study
* Survived until hospital discharge

Exclusion Criteria:

* Does not understand or speak English
* Has no fixed address
* Pre-existing cognitive impairment that prevents completion of the study assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who were enrolled in the ALTA, EDEN, OMEGA, or SAILS study.
Sampling Method: Non-Probability Sample
Enrollment: 922 (Actual)
Dates: Start 2007-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Individual Physical Function and Mental Health domains from SF-36 (for participants who complete the phone surveys); 6-minute walk distance and memory evaluation (for participants who attend the study visits) | Measured at Months 6 and 12

SECONDARY OUTCOMES:
Quality of life, mental health, memory and cognition, physical functioning, fatigue, walking ability, lung function, muscle strength, weight, dietary changes, and changes in muscle and fat composition | Measured at Months 6 and 12
  Short Form-36 domains, EQ-5D, Hospital Anxiety and Depression Scale, Impact of Event Scale-Revised, Mini-Mental State Examination, FACIT-Fatigue, Functional Performance Inventory, Wechsler Memory Scale - Logical Memory 1/2, Wechsler Adult Intelligence Scale - Digit Span and Similarities, Controlled Oral Word Association Test, Hayling Sentence Completion, Cognistat - Orientation and Judgment, Timed 4 Meter Walk, Hand grip, Manual Muscle Test, Maximal Inspiratory Pressure, Anthropometrics, DEXA

OTHER OUTCOMES:
Health Care Utilization, Employment Status, Health Insurance Status | Measured at Months 6 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Dale M. Needham, MD, PhD, Principal Investigator — Johns Hopkins University; Ramona O Hopkins, PhD, Principal Investigator — Intermountain Medical Center
Locations (6):
- United States (6):
  - University of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Wake Forest University, Winston-Salem, North Carolina
  - Vanderbilt University, Nashville, Tennessee
  - Intermountain Medical Center, Murray, Utah
  - University of Washington/Harborview Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Brown SM, Wilson E, Presson AP, Zhang C, Dinglas VD, Greene T, Hopkins RO, Needham DM; with the National Institutes of Health NHLBI ARDS Network. Predictors of 6-month health utility outcomes in survivors of acute respiratory distress syndrome. Thorax. 2017 Apr;72(4):311-317. doi: 10.1136/thoraxjnl-2016-208560. Epub 2016 Jul 20. PMID 27440140
- [Derived] Dinglas VD, Hopkins RO, Wozniak AW, Hough CL, Morris PE, Jackson JC, Mendez-Tellez PA, Bienvenu OJ, Ely EW, Colantuoni E, Needham DM. One-year outcomes of rosuvastatin versus placebo in sepsis-associated acute respiratory distress syndrome: prospective follow-up of SAILS randomised trial. Thorax. 2016 May;71(5):401-10. doi: 10.1136/thoraxjnl-2015-208017. Epub 2016 Mar 2. PMID 26936876
- [Derived] Needham DM, Colantuoni E, Dinglas VD, Hough CL, Wozniak AW, Jackson JC, Morris PE, Mendez-Tellez PA, Ely EW, Hopkins RO. Rosuvastatin versus placebo for delirium in intensive care and subsequent cognitive impairment in patients with sepsis-associated acute respiratory distress syndrome: an ancillary study to a randomised controlled trial. Lancet Respir Med. 2016 Mar;4(3):203-12. doi: 10.1016/S2213-2600(16)00005-9. Epub 2016 Jan 29. PMID 26832963
- [Derived] Dinglas VD, Huang M, Sepulveda KA, Pinedo M, Hopkins RO, Colantuoni E, Needham DM; NIH NHLBI ARDS Network. Personalized contact strategies and predictors of time to survey completion: analysis of two sequential randomized trials. BMC Med Res Methodol. 2015 Jan 9;15:5. doi: 10.1186/1471-2288-15-5. PMID 25575599
- [Derived] Needham DM, Dinglas VD, Bienvenu OJ, Colantuoni E, Wozniak AW, Rice TW, Hopkins RO; NIH NHLBI ARDS Network. One year outcomes in patients with acute lung injury randomised to initial trophic or full enteral feeding: prospective follow-up of EDEN randomised trial. BMJ. 2013 Mar 19;346:f1532. doi: 10.1136/bmj.f1532. PMID 23512759